CLINICAL TRIAL: NCT06707246
Title: A Randomized Clinical Trial Comparing the Efficacy and Safety of Secukinumab with Tofacitinib in the Treatment of Moderate to Severe Hidradenitis Suppurativa in Chinese Patients
Brief Title: A Randomized Trial Comparing the Efficacy and Safety of Secukinumab with Tofacitinib in the Treatment of Moderate to Severe Hidradenitis Suppurativa in Chinese Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Jinhua Central Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Ningbo No. 1 Hospital (Other); The First People's Hospital of Huzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0358
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; secukinumab; tofacitinib
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Secukinumab treatment group (Experimental): Participants will take secukinumab 300mg every week in the first month and every four weeks thereafter till 1 year
  Interventions: Drug: Secukinumab 300 MG; Tofacitinib 11mg
- Tofacitinib treatment group (Experimental): Participants will take tofacitinib 11mg daily for 1 year
  Interventions: Drug: Secukinumab 300 MG; Tofacitinib 11mg

INTERVENTIONS:
Drug: Secukinumab 300 MG; Tofacitinib 11mg — Tofacitinib tablet 11mg per tablet; Secukinumab 150mg/ml

SUMMARY:
The goal of this clinical trial is to compare the efficacy secukimumab versus tofacitinib in patients with moderate to severe hidradenitis suppurativa (HS)in adults. It will also learn about the safety of secukimumab and tofacitinib. The main questions it aims to answer are:

* Which treatment is more effective in patients with moderate to severe HS?
* What medical problems do participants have when taking secukimumab versus tofacitinib? Researchers will compare secukimumab versus tofacitinib to see which treatment works better to treat moderate to severe HS.

Participants will:

* Half of participants will take secukimumab every week in the first month and every four weeks thereafter till 1 year
* Another half of participants will take tofacitinib a tablet daily for 1 year
* Visit the clinic once every 2 weeks for checkups and tests in the first month, and every 4 weeks thereafter
* Keep a diary of their symptoms and the number of times they use a rescue inhaler

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participated in the study and signed informed consent.
* male and female subjects aged ≥18 years old (when signing the informed consent);
* Moderate to severe hidradenitis suppurativa: Hurley stage II or III.
* Patients voluntarily participated in the study and signed informed consent.
* male and female subjects aged ≥18 years old (when signing the informed consent);
* Moderate to severe hidradenitis suppurativa: Hurley stage II or III.
* Participants had stable disease at screening and baseline, with lesions located in ≥2 anatomical areas (≥1 at Hurley stage II/III), a total of ≥3 abscesses and inflammatory nodules (AN), and C-reactive protein levels > 3.0 mg/L.
* Participants had to have an intolerance, contraindication, or inadequate response to ≥3 months of oral antibiotic treatment for HS or relapse after discontinuation of treatment.
* Informed consents were signed according to the spirit of the Declaration of Helsinki.
* agree to receive regular treatment, follow-up, and relevant laboratory examinations in accordance with the clinical research protocol.

Exclusion Criteria:

* Allergy to drugs or excipients;
* patients who had previously used cubitumumab or tofacitinib;
* At the time of screening, the medical history, symptoms and examination results of the subjects suggested that the patients had active tuberculosis, active hepatitis B (HBV DNA> lower limit), hepatitis C, syphilis (TPPA+ but excluding active syphilis negative) or AIDS.
* any active malignant tumor or history of malignant tumor within 5 years, except cured skin squamous cell carcinoma or basal cell carcinoma or cervical cancer in situ;
* Severe infection or systemic infection requiring intravenous anti-infection therapy or hospitalization due to infection within 4 weeks before baseline;
* Severe, progressive or uncontrolled liver disease, defined as AST or ALT elevation > 3 times, or total bilirubin ULN elevation >2 times, which can be rescreened after treatment;
* Baseline drainage tube count > 20, diagnosis of inflammatory diseases other than HS, and history of chronic or recurrent infection or malignant tumor;
* history of drug abuse, attempted suicide or mental illness;
* those who participated in other clinical trials in the past 3 months;
* pregnant, breastfeeding, or planning to become pregnant during the trial;
* other conditions that the investigators thought should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Clinical response of HiSCR at week 12 week | Week 12
  abscess and inflammatory nodules with at least a 50% reduction in abscess from baseline, and no increase in drain fistula count relative to baseline

SECONDARY OUTCOMES:
Frequency and severity of adverse events (AE) and serious adverse events (SAE) | through study completion, usually 1 year
  Frequency and severity of AE and SAE throughout the study
Clinical response of HiSCR at week 52 week | 1 year
  abscess and inflammatory nodules with at least a 50% reduction in abscess from baseline, and no increase in drain fistula count relative to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Jiaqi Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No